CLINICAL TRIAL: NCT01013935
Title: A Spanish-Language Intervention to Enhance Routine HIV Patient Care Delivery [CARE+ Spanish]
Acronym: CARE+ Spanish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1RC1MH088307 (NIH)
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
Keywords: HIV treatment; ART adherence; Using new technology to improve adherence; CARE+; HIV-1 viral loads
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Full CARE+ Spanish computer-counseling group (Active Comparator)
  Interventions: Other: CARE+ Spanish computer counseling session
- Brief risk assessment study group only (control) (Active Comparator)
  Interventions: Other: CARE+ Spanish brief computer risk assessment session

INTERVENTIONS:
Other: CARE+ Spanish computer counseling session — The computer will ask patients questions about taking HIV medicine. The computer will also ask patients questions about sexual and substance use activities. The computer will let patients look at short videos on various HIV medicine and HIV risk reduction topics and will then help patients create a health plan. Patients will get an anonymous print out at the end of the session and can choose to share with health care provider. There are questions about depression, suicide, or domestic violence. If a patient's answers indicate that they may be depressed, suicidal, or currently in an abusive relationship, we will refer them to a health worker at the clinic. We will repeat the session every 3 months up to 12 months total.
  Other Names: CARE+
  Arms: Full CARE+ Spanish computer-counseling group
Other: CARE+ Spanish brief computer risk assessment session — The computer will ask patients questions about taking HIV medicine. The computer will also ask patients questions about sexual and substance use activities. We will repeat the session every 3 months up to 12 months total.
  Other Names: CARE+
  Arms: Brief risk assessment study group only (control)

SUMMARY:
The purpose of this study is to see if a computer counseling tool helps Spanish-speaking people living with HIV to have safer sex and to do well on their HIV medicines.

DETAILED DESCRIPTION:
Latinos are the fastest-growing group with some of the largest health disparities including HIV. Barriers including language are associated with lower antiretroviral therapy (ART) adherence seen among Latinos. There are no evidence-based interventions (randomized trials that significantly reduced viral load and HIV transmission risk to sexual partners - 'positive prevention') delivered in Spanish in routine clinical practice. Our computerized counseling tool (CARE+) in a phase III trial of English-speaking adults increased ART adherence and reduced viral load and condom use errors. We now propose a longitudinal effectiveness (phase IV) study to evaluate the impact of computerized counseling in audio-narrated Spanish in a busy urban HIV clinic. This 'CARE+ Spanish' proposal is responsive to 06-OD(OBSSR)-101, for new technologies to improve adherence in clinical practice. Aim 1: Adapt CARE+ Spanish for use during routine clinical visits by Spanish-speaking HIV clinic attendees using an expert panel to shorten content and add Spanish audio dialects; do usability testing (n≤8). Aim 2: Establish real-world utility of 'CARE+ Spanish'. Peer staff will recruit Spanish-speaking adults on ART who will be randomly assigned to intervention (Group A n=250) or risk-assessment control (B, n=250) for 0,3-,6-,9-month sessions; at 12-month session groups will switch to opposite arm (delayed intervention design). Linear and generalized linear mixed effects models will analyze impact on 30-day ART adherence, clinic visit adherence, HIV-1 viral load and sexual risks, and to assess whether any Group A changes are sustained at month 12, among an expected n=400 retained study participants (120 female, 280 male). Aim 3: Explore cultural acceptability of tool among clients and clinic providers. Conduct qualitative exit interviews with patients (n=75) to assess technology uptake factors, cultural/linguistic acceptability, and suggestions for ongoing use among older vs. younger, and US-born vs. foreign-born Latino groups. Conduct two focus groups with providers (n≤30) to assess perceived technology barriers/facilitators. Analysis will identify factors affecting acceptability, utilization, and impact. Technology tools like CARE+ present significant opportunities to bridge the health promotion delivery gap, especially if linguistically adapted for often-neglected groups such as Latinos (15% of the US population).

ELIGIBILITY:
Inclusion Criteria:

* Hispanic birth or ancestry
* Speaks Spanish (mono- or multi-lingual)

Exclusion Criteria:

* Lack of fluency in Spanish
* Thought disorder that precludes participation
* Inability to give informed consent due to altered mentation at time of enrollment (e.g., visibly inebriated or high).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
ART adherence | Every 3 months up to 12 months
HIV-1 viral load | Every 3 months up to 12 months
Sexual risks | Every 3 months up to 12 months
Clinic visit adherence | Every 3 months up to 12 months

SECONDARY OUTCOMES:
Qualitative exit interviews with patients (n=75) to assess technology uptake factors, cultural/linguistic acceptability, and suggestions for ongoing use among older vs. younger, and US-born vs. foreign-born Latino groups | At end of study
Two focus groups with providers (n≤30) to assess perceived technology barriers/facilitators | End of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ann Kurth, PhD, Principal Investigator — NYU
Locations (1):
- St. Luke's Roosevelt, New York, New York, United States

REFERENCES:
- [Derived] Kurth AE, Chhun N, Cleland CM, Crespo-Fierro M, Pares-Avila JA, Lizcano JA, Norman RG, Shedlin MG, Johnston BE, Sharp VL. Linguistic and Cultural Adaptation of a Computer-Based Counseling Program (CARE+ Spanish) to Support HIV Treatment Adherence and Risk Reduction for People Living With HIV/AIDS: A Randomized Controlled Trial. J Med Internet Res. 2016 Jul 13;18(7):e195. doi: 10.2196/jmir.5830. PMID 27417531